CLINICAL TRIAL: NCT04098991
Title: Improving White Matter Integrity With Thyroid Hormone
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Olusola Alade Ajilore, Associate Professor Associate Director, Residency Training and Education Co-Director, Adult/Neuroscience Research Track, University of Illinois at Chicago
Other Study IDs: 2016-0678; 5R21NS095723 (NIH)
Record Dates: First submitted 2018-02-27; First posted 2019-09-23 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Hypothyroidism
Keywords: neuroimaging; thyroid; white matter
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with primary hypothyroidism: All participants will receive the same treatment (levothyroxine, a synthetic T4 hormone replacement) at a dose that will be titrated using serum thyrotropin (TSH) levels as a goal, according to the American Thyroid Association Task Force recommendations
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — All participants will be treated for their hypothyroidism according to the standard of care as reflected in recent guidelines from the American Thyroid Association.

SUMMARY:
Animal studies have shown that thyroid hormone can improve white matter integrity after damage to myelin, which insulates and protects nerves. It is currently unknown whether this type of repair can occur in humans. The purpose of the proposed study is to examine the impact of thyroid hormone on white matter integrity in humans using two complementary, state-of-the-art neuroimaging techniques: high angular diffusion imaging and multicomponent relaxometry.

DETAILED DESCRIPTION:
The ability to promote and support remyelination has wide-ranging implications for a number of neuropsychiatric conditions from multiple sclerosis to major depression. Pre-clinical evidence has demonstrated that thyroid hormone treatment, in the form of triiodothyronine (T3) or tetraiodothyronine (T4), can promote and support remyelination by increasing myelin basic protein mRNA and protein, oligodendrocyte proliferation and maturation, and fractional anisotropy (a diffusion imaging measure of white matter integrity). Pilot data from the investigator's studies suggest that baseline thyroid status is correlated with the integrity of white matter tracts associated with major depression. To date, the impact of thyroid hormone administration on white matter tracts has not been studied in vivo in adult humans. The purpose of the proposed pilot study is to examine changes in white matter tract integrity using high angular diffusion imaging and multi-component relaxometry in a population of subjects clinically indicated to receive thyroid hormone for hypothyroidism. The investigators will scan patients with hypothyroidism at the initiation of treatment and at three and six months after starting thyroid hormone treatment. The investigators will also administer scales assessing mood and cognition which have been shown to correlate with white matter integrity. The investigators hypothesize that thyroid hormone treatment will be associated with an increase in fractional anisotropy, a decrease in radial diffusivity, and an increase in the myelin water fraction (markers of improved myelination) that will correlate with improvements in cognition and mood ratings. If successful, this will be the first demonstration of improved white matter integrity with thyroid hormone replacement and pave the way for therapies designed to restore structural brain connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-60 years of age
* A diagnosis of primary hypothyroidism from autoimmune thyroiditis (Hashimoto)
* Able to give informed consent.

Exclusion Criteria:

* Major depressive disorder with or without active suicidal ideation
* Mild or major neurocognitive disorder;
* Presence of contraindications to magnetic resonance imaging (presence of ferrous-containing metals within the body (e.g., aneurysm clips, shrapnel/retained particles)
* Inability to tolerate small, enclosed spaces without anxiety (e.g., claustrophobia)
* Unwilling/unable to sign informed consent document
* Positive urine drug screen results;
* Pregnancy (positive pregnancy test), trying to become pregnant, or lactation

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We are seeking a population of subjects clinically indicated to receive thyroid hormone for hypothyroidism.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
High Angular Diffusion Tensor Imaging | 6 months
  Change in baseline white matter track integrity at 3 months and 6 months
Multi-Component Relaxometry | 6 months
  Change in baseline white matter track integrity at 3 months and 6 months

SECONDARY OUTCOMES:
Patient Health Questionaire | Collected at Baseline, 3 month follow-up, 6 month follow-up
  Self-report measure of depression severity, Items are summed (Not at all = 0; Several days = 1; More than half the days = 2; Nearly every day = 3), yielding a score from 0 to 27
NIH Toolbox : Dimensional Change Card Sort Test | Collected at Baseline, 3 month follow-up, 6 month follow-up
  Behavioral measures of executive functioning
NIH Toolbox : Pattern Comparison Processing Speed Test | Collected at Baseline, 3 month follow-up, 6 month follow-up
  Behavioral measures of processing-speed measure
NIH Toolbox : Flanker Inhibitory Control and Attention Test | Collected at Baseline, 3 month follow-up, 6 month follow-up
  Behavioral measures of attention

CONTACTS AND LOCATIONS:
Overall Officials: Olusola A Ajilore, MD/PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04098991/Prot_SAP_000.pdf